CLINICAL TRIAL: NCT00280436
Title: A Randomized, Double-blind, Placebo-controlled, Cross-over Study to Evaluate the Effects of GW679769 on Polysomnographic Sleep Recordings, Subjective Sleep Assessment, and Daytime Cognitive Function in Elderly and Non-elderly Subjects With Primary Insomnia
Brief Title: Effects Of GW679769 On Sleep Onset And Maintenance,And Next Day Functioning In The Elderly And Non-elderly With Primary Insomnia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MAD105514
Record Dates: First submitted 2006-01-19; First posted 2006-01-23 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Sleep Initiation and Maintenance Disorders; Insomnia
Keywords: Polysomnography; Electroencephalography; Primary Insomnia; Cognition; Sleep
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — casopitant

INTERVENTIONS:
Drug: GW679769

SUMMARY:
This study is designed to find the optimal (best) doses of GW679769 that promote sleep onset and maintain sleep during two consecutive nights of dosing without significant next-day thinking impairment and drowsiness in subjects with primary insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Difficulty going to sleep and/or staying asleep for at least the past 3 months.
* Insomnia must result in significant distress or impairment in functioning at home, socially or at work.
* Otherwise good health with no significant or unstable medical disorder including psychiatric, neurological, endocrine, heart, lung or gastrointestinal disorders, drug/alcohol abuse, cognitive impairment, cancer or chronic pain conditions such as arthritis.

Exclusion Criteria:

* History of other sleep disorders such as sleep apnea or restless leg syndrome.
* Regular sleep habits, including bedtime between 9 PM and midnight.
* Nightshift/rotating shift work, frequent napping or planned travel across >2 time zones.
* Use to moderate use of nicotine, caffeine and alcoholic products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2006-01; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Comparison of GW679769 and placebo on the average time needed to fall asleep after bedtime dosing on two consecutive nights, as assessed by electroencephalography and other physiological changes during sleep. | 48 Hours

SECONDARY OUTCOMES:
Comparison of GW679769 and placebo on sleep maintenance and duration after bedtime dosing on two consecutive nights, as assessed by electroencephalography and subject diaries, and on next-day memory, alertness and physical coordination. | 48 Hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (24):
- United States (24):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Glendale, California
  - GSK Investigational Site, Redlands, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Brandon, Florida
  - GSK Investigational Site, Kissimmee, Florida
  - GSK Investigational Site, Naples, Florida
  - GSK Investigational Site, Spring Hill, Florida
  - GSK Investigational Site, Austell, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Northfield, Illinois
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Chevy Chase, Maryland
  - GSK Investigational Site, Frederick, Maryland
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Lafayette Hill, Pennsylvania
  - GSK Investigational Site, Warwick, Rhode Island
  - GSK Investigational Site, Anderson, South Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Fairfax, Virginia